CLINICAL TRIAL: NCT03759743
Title: a Randomised, Double Blind, Placebo Controlled Study to Evaluate the Efficacy and Safety of LMT1-48 on Reducing Body Fat in Overweight Subject
Brief Title: Evaluate the Efficacy and Safety of LMT1-48 on Reducing Body Fat in Overweight Subject
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT13-KR17OWT712
Record Dates: First submitted 2018-11-14; First posted 2018-11-30 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental)
  Interventions: Dietary Supplement: LMT1-48
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: LMT1-48 — capsules containing Probiotics
  Arms: Probiotics
Dietary Supplement: Placebo — capsules that did not contain any probiotics
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of LMT1-48(Probiotics) compared to a placebo in reducing the body fat in overweight subjects

ELIGIBILITY:
Inclusion Criteria:

* Age between 19 and 70 years
* Overweight (25 kg/m2 ≤ body mass index (BMI) < 30 kg/m2)

Exclusion Criteria:

* Pregnancy or breast-feeding
* Unstable body weight (body weight change > 10% within 3 months before screening)

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2019-08-17 (Actual); Study Completion 2020-01-07 (Actual)

PRIMARY OUTCOMES:
change from baseline fat percentage at 12 week | at baseline and 12-week follow-up
  the body composition of the subjects was measured via dual-energy X-ray absorptiometry (DEXA) to determine

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, South Korea

REFERENCES:
- [Derived] Sohn M, Jung H, Lee WS, Kim TH, Lim S. Effect of Lactobacillus plantarum LMT1-48 on Body Fat in Overweight Subjects: A Randomized, Double-Blind, Placebo-Controlled Trial. Diabetes Metab J. 2023 Jan;47(1):92-103. doi: 10.4093/dmj.2021.0370. Epub 2022 Apr 29. PMID 35487505